CLINICAL TRIAL: NCT06962228
Title: A Multicenter Observational Cross-sectional Clinical Trial of Cross-cultural Adaptation of the Chinese Version of QoLAF-Q (Quality of Life in Patients With Anal Fistula Questionnaire)
Brief Title: Cross-cultural Adaptation of the Chinese Version of QoLAF-Q (Quality of Life in Patients With Anal Fistula Questionnaire) ：A Multi-center Study
Status: Not yet recruiting | Type: Observational
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Wei Zhang, Director of the department of colorectal surgery, Changhai Hospital
Other Study IDs: QoLAF-Q
Record Dates: First submitted 2025-04-22; First posted 2025-05-08 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-04

CONDITIONS: Anal Fistula
MeSH Terms: conditions — Rectal Fistula

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- anal fistula patients
  Interventions: Procedure: Anal fistula surgery

INTERVENTIONS:
Procedure: Anal fistula surgery — Anal fistula incision, anal fistula excision, anal fistula hanging

SUMMARY:
The investigators verify the reliability and practicality of the Chinese adaptation results of QoLAF-Q, which helps Chinese doctors better master the methods and techniques of quality of life assessment.

DETAILED DESCRIPTION:
When the investigators conduct cross-cultural adaptation to verify the applicability of QoLAF-Q in China, the investigators also compare it with the cross-cultural adaptation results of other language versions of this scale. While verifying the reliability and practicality of the Chinese adaptation results of QoLAF-Q, the investigators also explore its differences, which helps Chinese doctors better master the methods and techniques of quality of life assessment, pay more attention to the physical and mental health of patients, improve the quality of life and satisfaction of patients, and provide a reference for the development of more scientific, effective, and practical scales.

ELIGIBILITY:
Inclusion Criteria:

1. meeting the diagnostic criteria for anal fistula in the "Diagnostic Criteria for Anal Fistula (2004 Edition)", and being diagnosed through clinical examinations, digital rectal examinations, anorectal ultrasound, MRI, and other examinations;
2. being 18 years old or above;
3. having clear consciousness and being able to understand and cooperate to complete the questionnaire survey;
4. voluntarily signing the informed consent form.

Exclusion Criteria:

1. having other serious anorectal diseases, such as anal fissure, rectal prolapse, colorectal cancer, etc.;
2. having severe dysfunction of important organs such as the heart, liver, and kidneys;
3. suffering from mental diseases or having cognitive impairments;
4. having undergone anorectal surgery or other major surgeries that may affect the quality of life recently (within 3 months).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: anal fistula patients who visited the anorectal surgery wards and outpatient departments of tertiary hospitals across the country
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Cronbach's α coefficient | immediately after filling out the questionnaires
  Reliability analysis was used to study the reliability and precision of the responses to quantitative data (especially the attitude scale questions).The Cronbach's α coefficient is a commonly used reliability index, which measures the correlation between various items in the scale and determines whether each item in the scale is measuring the same concept or trait. If the Cronbach's alpha coefficient is high, it indicates that the correlation among the items is strong, and the internal consistency of the scale is good, meaning that these items can relatively consistently reflect the psychological trait or concept being measured.In the reliability analysis of this study, if the Cronbach's α coefficient reaches above 0.8, it indicates that each item can effectively revolve around the core concept of "the quality of life of patients with anal fistula", and there is a high degree of consistency among these items.

SECONDARY OUTCOMES:
KMO value | immediately after filling out the questionnaires
  Validity analysis is used to study the rationality of the design of quantitative data (especially items in attitude scales). For the validity analysis of this scale, it is required to use the KMO value to determine whether the data obtained after converting the subjective choices of patients into Likert scale scores are reasonable and whether they can be used for factor analysis, so as to judge the appropriateness of information extraction and verify the validity level of the data.
Factor analysis of QoLAF-Q(quality of life in patients with anal fistula questionnaire) | immediately after filling out the questionnaires
  The factor analysis of the Quality of Life in Anal Fistula Questionnaire (QoLAF-Q) is used to verify the applicability of QoLAF-Q in China through cross-cultural research, which includes two parts: exploratory factor analysis(EFA) and confirmatory factor analysis(CFA). EFA extracts the latent factors in the scale through methods such as principal component analysis to determine the structural dimensions of the scale.Based on EFA, CFA uses structural equation modeling to verify the structure of the scale and further evaluate the construct validity of the scale. By comparing the model fit indices, such as the chi-square to degrees of freedom ratio (χ²/df), goodness-of-fit index (GFI), etc, the degree of fit between the model and the data is judged.When the various indicators in the factor analysis of QoLAF-Q are basically higher than the predicted values, it indicates that the QoLAF has good applicability for the assessment of Chinese patients.

IPD SHARING:
Plan to Share IPD: No